CLINICAL TRIAL: NCT02369926
Title: Phase 2a, Randomized, Double-Blind, Placebo Controlled, Parallel Group Study of the Safety, Tolerability, and Proof-of-Concept Efficacy of Lisinopril in Patients With Relapsing-Remitting Multiple Sclerosis (RRMS), Stage 1
Brief Title: Endpoint Calibration for a Phase 2 Study of Lisinopril in Multiple Sclerosis
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Transparency Life Sciences (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Health Services Research
Other Study IDs: TLS-002
Record Dates: First submitted 2015-02-10; First posted 2015-02-24 (Estimated); Last update posted 2017-10-12 (Actual); Status verified 2017-10

CONDITIONS: Multiple Sclerosis, Relapsing-Remitting
Keywords: multiple sclerosis; telemedicine; remote monitoring; lisinopril
MeSH Terms: conditions — Multiple Sclerosis, Relapsing-Remitting; Multiple Sclerosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Group 1 (Active Comparator): Participants will be separated into two groups for scheduling purposes. Each group will complete the Multiple Sclerosis Functional Composite (MSFC) once weekly at the study site and once weekly at home for three weeks. They will alternate their visit dates with Group 2.
  Interventions: Procedure: Multiple Sclerosis Functional Composite; Procedure: Mobile Multiple Sclerosis Functional Composite
- Group 2 (Active Comparator): Participants will be separated into two groups for scheduling purposes. Each group will complete the Multiple Sclerosis Functional Composite (MSFC) once weekly at the study site and once weekly at home for three weeks. They will alternate their visit dates with Group 1.
  Interventions: Procedure: Multiple Sclerosis Functional Composite; Procedure: Mobile Multiple Sclerosis Functional Composite

INTERVENTIONS:
Procedure: Multiple Sclerosis Functional Composite — The MSFC is a diagnostic test that measures multiple sclerosis symptoms. It includes a timed walk test, 9-hole peg test, and paced auditory serial addition test. The MSFC is administered in-person at the study site.
  Other Names: MSFC
Procedure: Mobile Multiple Sclerosis Functional Composite — The mMSFC is a diagnostic test that measures multiple sclerosis symptoms from. It includes a timed walk test, 9-hole peg test, and paced auditory serial addition test. All aspects of this exam are completed from a participant's home using remote sensing technology and video conferencing.
  Other Names: mMSFC

SUMMARY:
This study aims to calibrate the Multiple Sclerosis Functional Composite (MSFC) for home implementation in a phase 2 trial of lisinopril in multiple sclerosis. In this initial stage, participants are required to travel to the study site one day a week for three weeks to complete the MSFC. They are also required to complete the MSFC at home once weekly for three weeks using remote sensing technology and video conferencing.

ELIGIBILITY:
Inclusion Criteria:

1. Males and females between the ages of 18 and 64.
2. Documented informed consent
3. Documented diagnosis of RRMS via 2010 McDonald Criteria
4. Normal blood pressure at baseline: 90-140 mmHg systolic AND 60-90 mmHg diastolic
5. Baseline score of 0-5.5 on Kurtzke's Expanded Disability Status Scale (EDSS)
6. Availability of a person in the home who is physically able and willing to steady the subject if s/he loses balance during the walk test.

Exclusion Criteria:

1. Hypotensive at baseline: <90 mmHg systolic or <60 mmHg diastolic
2. Hypertensive at baseline: >140 mmHg systolic or >90 mmHg diastolic
3. Bradycardia at baseline: < 50 bpm

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2014-11; Primary Completion 2018-06 (Estimated)

PRIMARY OUTCOMES:
Safety of mMSFC Tally | Week 6
  Safety of remote video administration of the mMSFC will be calculated at the end of the study by calculating and comparing the instances of balance-related safety issues.
MSFC Score Comparison | Week 6
  mMSFC scores will be compared to MSFC scores for proof of calibration.
Mobile Timed Walk Test Value Comparison | Week 6
  Mobile timed walk times will be compared to 25-foot timed walk test times for proof of calibration.
Mobile 9-hole Peg Test Time Comparison | Week 6
  Mobile 9HPT time will be compared to 9 HPT time for proof of calibration.
Mobile Paced Auditory Serial Addition Test Score Comparison | Week 6
  Mobile PASAT3 scores will be compared to PASAT3 scores for proof of calibration.

CONTACTS AND LOCATIONS:
Overall Officials: Tomasz Sablinski, MD, PhD, Study Director — Transparency Life Sciences
Locations (1):
- Icahn School of Medicine at Mount Sinai, New York, New York, United States